CLINICAL TRIAL: NCT04956367
Title: Efficacy of Ablative Fractional Carbon Dioxide Laser Combined With Autologous Platelet-rich Plasma Versus Ablative Fractional Carbon Dioxide Laser and Placebo in the Treatment of Striae Gravidarum: a Randomized Clinical Trial
Brief Title: Efficacy of Fractional Carbon Dioxide Laser Combined With Platelet-rich Plasma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jose R. Reyes Memorial Medical Center (Other Government)
Responsible Party: Principal Investigator, Ivan Arni Preclaro, Efficacy of ablative fractional carbon dioxide laser combined with autologous platelet-rich plasma versus ablative fractional carbon dioxide laser and placebo in the treatment of striae gravidarum: a randomized clinical trial, Jose R. Reyes Memorial Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-054
Record Dates: First submitted 2021-06-22; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Striae Gravidarum
Keywords: Striae Gravidarum; carbon dioxide laser; platelet-rich plasma
MeSH Terms: conditions — Striae Distensae | interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Used a computer-generated software to randomize the area to be treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CO2 laser with PRP (Experimental): After anesthetizing the area and undergo one pass of ablative fractional CO2 laser (Smaxel, iDS, Korea) using the following settings: energy = 50 mJ; pulse duration = 2 ms; and density level = 15, PRP will be injected through nappage technique at 1 cm intervals for three treatment sessions at four-week intervals.
  Interventions: Procedure: Ablative fractional carbon dioxide laser combined with autologous platelet-rich plasma; Device: CO2 laser with PRP
- CO2 laser with placebo (Placebo Comparator): After anesthetizing the area and undergo one pass of ablative fractional CO2 laser (Smaxel, iDS, Korea) using the following settings: energy = 50 mJ; pulse duration = 2 ms; and density level = 15, pNSS will be injected through nappage technique at 1 cm intervals for three treatment sessions at four-week intervals.
  Interventions: Procedure: Ablative fractional carbon dioxide laser combined with autologous platelet-rich plasma; Device: CO2 laser with placebo

INTERVENTIONS:
Procedure: Ablative fractional carbon dioxide laser combined with autologous platelet-rich plasma — Carbon dioxide laser (Smaxel.878.4810) was FDA-approved device used in dermatology practice. PRP was described as having growth factors to be used to promote healing.
Device: CO2 laser with PRP — CO2 laser with PRP
  Arms: CO2 laser with PRP
Device: CO2 laser with placebo — CO2 laser with placebo
  Arms: CO2 laser with placebo

SUMMARY:
This study determined the efficacy of ablative fractional carbon dioxide laser combined with autologous platelet-rich plasma versus ablative fractional carbon dioxide laser with placebo in the treatment of striae gravidarum of postpartum Filipino women.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum patients with ages 18 to 45 years
* Fitzpatrick skin type III-V
* having bilateral symmetrical SG of red, white or a combination of both types.

Exclusion Criteria:

* pregnancy
* breastfeeding
* heavy consumption of alcoholic beverages
* dermatological conditions such as psoriasis, systemic lupus erythematosus and atopic dermatitis
* uncontrolled hypertension, diabetes mellitus, heart disease, acute and chronic liver/kidney impairment/disease;
* elevated liver function tests (SGPT, SGOT), and serum creatinine;
* intake of any medications that may influence the outcome of the study;
* intake of any vitamins/minerals or any supplements in the past 6 months; and
* application of any topical agents (e.g., whitening, anti-aging) in the past 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 16 weeks
  Change in appearance based from clinical photos done in baseline, week 6, week 10, week 14 and week 16 . This will be assessed by quartile grading scale (poor, <25% improvement; fair, 25-50% improvement; good, 51-75% improvement; and excellent, >75% improvement)

SECONDARY OUTCOMES:
Patient satisfaction rate | 16 weeks
  Self-reported by the patient using a quartile grading system with the following grades: 0 as poor; 1 as fair; 2 as satisfied; or 3 as very satisfied. The rating will be done at weeks 6, 10, 14 and 16.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Arni C Preclaro, MD, Principal Investigator — Jose R. Reyes Memorial Medical Center
Locations (1):
- Jose R Reyes Memorial Medical Center, Manila, NCR, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Faghihi G, Keyvan S, Asilian A, Nouraei S, Behfar S, Nilforoushzadeh MA. Efficacy of autologous platelet-rich plasma combined with fractional ablative carbon dioxide resurfacing laser in treatment of facial atrophic acne scars: A split-face randomized clinical trial. Indian J Dermatol Venereol Leprol. 2016 Mar-Apr;82(2):162-8. doi: 10.4103/0378-6323.174378. PMID 26924405